CLINICAL TRIAL: NCT05962320
Title: Effect of Enhanced Recovery After Surgery Protocol Based Care on Patient Outcomes in Children With Appendicitis: a Randomized Controlled Trial
Brief Title: Effect of Modified ERAS Protocol on Clinical Outcomes in Pediatric Patients With Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Buket MERAL, Research asistant - MSc, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KaradenizTU
Record Dates: First submitted 2023-06-18; First posted 2023-07-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: ERAS; Surgery; Appendicitis
Keywords: Appendectomy; Nurse; Child; Pain; Length of Stay; Anxiety; Fear; Vomiting
MeSH Terms: conditions — Appendicitis; Pain; Anxiety Disorders; Vomiting | interventions — Educational Status; Counseling; Drainage; Urinary Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mERAS Group (Experimental): * Education and counselling of patients and their parents
  * Avoiding the use of nasogastric catheters, drains and urinary catheters or/and removing them as early as possible
  * Stimulation of intestinal motility in the postoperative period
  * Initiation of oral intake in the early postoperative period
  * Early removal of the patient by reducing postoperative IV fluid infusion
  * Initiation of early mobilization of the patient in the postoperative period
  * Providing pain management with opioid-limiting pharmacologic and non-pharmacological interventions
  * Non-pharmacological interventions in management nausea and vomiting
  * Management of thirsty through non-pharmacological interventions
  * Management of fear and anxiety through non-pharmacological interventions
  Interventions: Other: Education and counselling; Other: Avoiding the use of nasogastric catheters, drains and urinary catheters; Other: Stimulation of intestinal motility in the postoperative period; Other: Initiation of oral intake in the early postoperative period; Other: Early removal of the patient by reducing postoperative IV fluid infusion; Other: Initiation of early mobilization of the patient in the postoperative period; Other: Reducing opioid use and ensuring pain management; Other: Implement nausea and vomiting prophylaxis; Other: Management of thirsty; Other: Management of fear and stress
- Standart Care Group (No Intervention): Patients in this group will receive standard care according to the practices of the clinic where the study will be conducted.

INTERVENTIONS:
Other: Education and counselling — Education and counselling of patients and their parents
  Arms: mERAS Group
Other: Avoiding the use of nasogastric catheters, drains and urinary catheters — Avoiding the use of nasogastric catheters, drains and urinary catheters or/and removing them as early as possible
  Arms: mERAS Group
Other: Stimulation of intestinal motility in the postoperative period — Stimulation of intestinal motility in the postoperative period
  Arms: mERAS Group
Other: Initiation of oral intake in the early postoperative period — Initiation of oral intake in the early postoperative period
  Arms: mERAS Group
Other: Early removal of the patient by reducing postoperative IV fluid infusion — Early removal of the patient by reducing postoperative IV fluid infusion
  Arms: mERAS Group
Other: Initiation of early mobilization of the patient in the postoperative period — Initiation of early mobilization of the patient in the postoperative period
  Arms: mERAS Group
Other: Reducing opioid use and ensuring pain management — Reducing opioid use and ensuring pain management
  Arms: mERAS Group
Other: Implement nausea and vomiting prophylaxis — Implement nausea and vomiting prophylaxis
  Arms: mERAS Group
Other: Management of thirsty — Management of thirsty
  Arms: mERAS Group
Other: Management of fear and stress — Use of recommended non-pharmacological interventions in the management of fear and stress
  Arms: mERAS Group

SUMMARY:
Acute appendicitis is the most common abdominal emergency with more than 15 million cases reported worldwide. Although appendectomy is considered a safe surgical procedure, the incidence of complications is up to 10%. The Enhanced Recovery After Surgery (ERAS) has developed guidelines to improve postoperative patient outcomes. The protocol, which consists of more than 20 interventions in the preoperative, intraoperative and postoperative periods, shows that early discharge can be possible with multidisciplinary care given to surgical patients without risking patient safety.

DETAILED DESCRIPTION:
Appendicitis is a common clinical condition and often requires emergency treatment. Although appendectomy is a safe surgical procedure, there is a risk of complications. Pain is common, especially in the postoperative period, and the lack of care management leads to delayed mobilization and oral intake, delayed recovery and prolonged length of hospital stay. However, pain, nausea-vomiting, thirst, fear and stress could be managed with perioperative care. In addition, it is reported that the care provided based on the ERAS protocol shortens the length of hospital stay. In this respect, the aim of this study was to investigate the effect of ERAS protocol-based care on the length of hospital stay of children who were planned to undergo appendectomy. Postoperative pain level, stress and fear level, time to first mobilization, flatulence, defecation and oral intake, nausea, thirst were the secondary outcomes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥6 years and ≤17 years, girls or boys
* Underwent appendectomy
* Written informed consent or requirements of local/national ethical committee

Exclusion Criteria:

* ASA (American Society of Anesthesiologists, ASA) score of ≥ 3
* Any comorbidity/contraindication that may prevent mobilization and oral feeding

The withdrawal criteria:

* During the surgery, the surgeon classified appendicitis as grade 0 (no appendicitis) or grade IIIB and above,
* during the postoperative period need for intensive care hospitalization patients in the control or the mERAS protocol group were staying in the same room,
* contraindications to the application of any intervention in the intervention group and/or the primary physician not approving the application of the intervention,
* the compliance rate of the interventions determined in the modified ERAS protocol being below 80%,
* the development of any other comorbidity (urinary calculi, intussusception, etc.),
* the change in the type of surgery during the operation, conversion from laparoscopic to open appendectomy.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Postoperative length of hospital stay | From the end of surgery until hospital discharge, up to 10 days
  The postoperative length of hospital stay will be calculated in hours. Higher scores indicate delayed discharge. This means a worse outcome.

SECONDARY OUTCOMES:
Complications | up to 30 days after discharge
  Postoperative minor and major complications will be recorded.
Readmission | up to 30 days after discharge
  Readmission to the hospital will be recorded in hours.
Postoperative pain | Assessed 5 times on the day of surgery (Postoperative Day 0) after patient awakening, approximately every 4-6 hours
  Postoperative pain will be evaluated with Numeric Pain Scale. Higher scores mean more severe pain, worse outcome
Postoperative fear | Assessed 2 times on the day of surgery (Postoperative Day 0) after patient awakening, approximately every 12 hours
  Postoperative fear will be evaluated with Children's Fear Scale. Higher scores mean more severe fear, worse outcome.
Postoperative anxiety | Assessed 2 times on the day of surgery (Postoperative Day 0) after patient awakening, approximately every 12 hours
  Postoperative anxiety will be evaluated with Children's State Anxiety. Higher scores mean more severe anxiety, worse outcome.
Postoperative nausea-vomiting | Assessed 5 times on the day of surgery (Postoperative Day 0) after patient awakening, approximately every 4-6 hours
  Postoperative nausea-vomiting will be evaluated with Baxter Retching Faces Scale. Higher scores mean more severe nause, worse outcome
Postoperative thirst | up to the first oral intake, an average 2 days
  Postoperative thirst will be evaluated with Numeric Thirst Scale. Higher scores mean more severe pain, worse outcome.
Time of first mobilization | up to the first mobilization, an average 12 hours
  The first time of postoperative mobilization will be recorded in hours. Higher scores indicate delayed mobilization. This means a worse outcome.
Time of first defecation | up to the first defecation, an average 3 days
  The first time of postoperative defecation will be recorded in hours. Higher scores indicate delayed defecation. This means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Buket MERAL, Msc, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data, with identifying information concealed, forming the basis of the results reported in this article, will be made available upon reasonable request to the corresponding author 6-12 months after publication of the article. Researchers should contact the corresponding author to request access to the data.